CLINICAL TRIAL: NCT02644850
Title: Comparison of Gated Blood-pool SPECT Using CZT Camera and Echocardiogram for Ventricular Ejection Fraction Estimation
Brief Title: Comparison of Gated Blood-pool SPECT and Echocardiogram for Ventricular Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201508081RINA
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare the calculated biventricular ejection fraction from cadmium-zinc-telluride (CZT) single photon emission computed tomography (SPECT) with planar equilibrium radionuclide angiography (ERNA), first-pass radionuclide ventriculography (FP-RNV) and echocardiogram.

DETAILED DESCRIPTION:
To evaluate the feasibility of using CZT SPECT as an "all-in-one" technique to provide information on both left ventricular ejection fraction (LVEF) and right ventricular ejection fraction (RVEF) derived from a single examination and compare with the values from traditional planar ERNA, FP-RNV and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent transthoracic echocardiogram and resting cardiac function within interval of 90 days of each other

Exclusion Criteria:

* Pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent transthoracic echocardiogram and resting cardiac function within interval of 90 days of each other
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Measure the biventricular ejection fraction | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Fang Cheng, M.D., Principal Investigator — National Taiwan University Hospital and National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital and National Taiwan University College of Medicine, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No